CLINICAL TRIAL: NCT05344378
Title: Refining and Implementing Technology-Enhanced Family Navigation to Promote Early Access and Engagement With Mental Health Services for Youth With Autism
Acronym: ATTAIN NAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Kaiser Permanente (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Nicole Stadnick, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 200147; 1R34MH120190-01A1 (NIH)
Record Dates: First submitted 2022-04-07; First posted 2022-04-25 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Autism Spectrum Disorder; Implementation Science; Mental Health; Behavioral Health
MeSH Terms: conditions — Autism Spectrum Disorder; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The investigators used a stepped wedge cluster randomized hybrid Type I effectiveness-implementation design to test the effects of technology-enhanced FN on service and clinical outcomes while gathering information on FN implementation (feasibility and acceptability). This design will also facilitate the early identification of technology enhancements that may require redesign to allow for testing of the redesigned enhancements during the subsequent step.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1 Month Baseline Period (No Intervention): Initial baseline period for rollout at 6 different clinics throughout the year-long intervention period using a step-wedge design.
- Stage 1 Enrollment (Experimental): Enrollment of 2 clinics over 4 months including 5 PCPs per clinic (2 total clinics).
  Interventions: Behavioral: ATTAIN NAV Technology-Enhanced Family Navigation Model
- Stage 2 Enrollment (Experimental): Addition of 2 clinics with modifications over 4 months including 5 PCPs per clinic (4 total clinics).
  Interventions: Behavioral: ATTAIN NAV Technology-Enhanced Family Navigation Model
- Stage 3 Enrollment (Experimental): Addition of 2 clinics with modifications over 4 months including 5 PCPs per clinic (4 total clinics).
  Interventions: Behavioral: ATTAIN NAV Technology-Enhanced Family Navigation Model

INTERVENTIONS:
Behavioral: ATTAIN NAV Technology-Enhanced Family Navigation Model — The purpose of ATTAIN NAV is to test the impact of family navigation in multiple primary care clinics in Southern California for children with autism who have additional mental health needs. Family navigation includes: screening and behavioral health referral, supporting access to behavioral health services, engaging in evidence-based treatment, monitoring to achieve family goals, family strengthening, and connecting to concrete resources.
  Arms: Stage 1 Enrollment; Stage 2 Enrollment; Stage 3 Enrollment

SUMMARY:
This project, Refining and Implementing Technology-Enhanced Family Navigation to Promote Early Access and Engagement with Mental Health Services for Youth with Autism (ATTAIN NAV) is focused on adapting and implementing family navigation in primary care settings to help accelerate and facilitate engagement in mental health and community services for children with autism and their families.

DETAILED DESCRIPTION:
Efficient and effective access to and engagement with evidence-based mental health (MH) services for children with autism spectrum disorder (ASD) is critically needed but requires a tailored approach. This project is critical in establishing integrated and sustainable local capacity to provide evidence-based MH care for children (ages 4-16 years) with ASD+ (i.e., children with ASD and co-occurring psychiatric disorders). Specifically, the overarching goal of this mixed methods proposal is to collaboratively adapt Family Navigation (FN) content, navigator activities and training for children with ASD+, identify and design technology enhancements to FN that will target key mechanisms to impact implementation, service and clinical outcomes, key interrelated outcomes for implementation research. The research team will leverage existing partnerships with primary care practices and lay health worker organizations in San Diego County to establish a community-academic partnership that will guide adaptations to FN for children with ASD+ (Aim 1), co-design of the navigator-facing technology enhancements (Aim 2) and trial the adapted and technology-enhanced FN (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Primary Care Providers

1. Employed as staff at participating primary care practice
2. Experience providing primary care to children with ASD
3. For Aim 3 only: Has at least five eligible children on current caseload

Inclusion Criteria for Child/Caregiver Participants (Aim 3 only)

1. Child age 4-16 years.
2. Child has a diagnosis of autism spectrum disorder documented in medical chart.
3. Child is receiving primary care at a participating primary care practice.
4. Child screens in the clinically significant range on the Pediatric Symptom Checklist at baseline.
5. Speaks English or Spanish.
6. Caregiver of an eligible child.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM) | Distributed at study completion, an average of 1 year.
  4-item questionnaire measure adapted for the ATTAIN NAV study to assess acceptability of the overall adapted FN intervention. Four-item measures of implementation outcomes that are considered indicators of implementation success. Response Scale: 1 = Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Completely agree. Scoring Instructions: Scales can be created for each measure by averaging responses. Scale values range from 1 to 5. No items need to be reverse coded. Higher scores indicate a better outcome.
Feasibility of Intervention Measure (FIM) | Distributed at study completion, an average of 1 year.
  4-item questionnaire measure adapted for the ATTAIN NAV study to assess feasibility of the overall adapted FN intervention. Four-item measures of implementation outcomes that are considered indicators of implementation success. Response Scale: 1 = Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Completely agree. Scoring Instructions: Scales can be created for each measure by averaging responses. Scale values range from 1 to 5. No items need to be reverse coded. Higher scores indicate a better outcome.
Appropriateness of Intervention Measure (AIM) | Distributed at study completion, an average of 1 year.
  4-item questionnaire measure adapted for the ATTAIN NAV study to assess appropriateness of the overall adapted FN intervention. Four-item measures of implementation outcomes that are considered indicators of implementation success. Response Scale: 1 = Completely disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Completely agree. Scoring Instructions: Scales can be created for each measure by averaging responses. Scale values range from 1 to 5. No items need to be reverse coded. Higher scores indicate a better outcome.
the Navigation Satisfaction Tool (NAVSAT) | Measured at the completion of family navigation services for each family, approximately 4 months after enrolling.
  22 item questionnaire assess satisfaction with the relationship with the navigator and with the referred services to which the navigator facilitated access. Response scale: 1= Extremely Dissatisfied 2=Dissatisfied 3=Fairly Dissatisfied 4= Not dissatisfied nor satisfied 5= Fairly Satisfied 6= Satisfied 7= Extremely Satisfied. Higher scores indicate a better outcome.
Navigator Fidelity | Measured at the completion of family navigation services for each family, approximately 4 months after enrolling.
  The investigators will adapt fidelity procedures (observational and self-report) from the navigator training curriculum used in MOST. Fidelity will be defined as demonstrating mastery on at least 80% of all components (e.g., navigator introduces purpose of navigation during initial contact, conducts assessment on barriers to attendance of first MH appointment). Fidelity will be measured at the completion of the navigator protocol for each family.
Eyberg Child Behavior Inventory (ECBI) | Measured at the start and completion of family navigation services for each family, approximately week 0 and 4 months after enrolling.
  The ECBI is a 36-item caregiver-report measure that assesses the frequency and intensity of child behavior problems. It has shown sensitivity to change over time. There are two scores: an Intensity score (frequency of behaviors) and a Problem (number of challenging behaviors) score. Both are converted into t-scores (M =50; SD=10). Scoring: on a 1-7 scale: How often does this occur with your child? ranging from (1) Never to (7) Always. There is a secondary scale that asks is this a problem for you? Yes/No.
Parent Activation Measure for Developmental Disabilities (PAM-DD) | Measured at the completion of family navigation services for each family, approximately 4 months after enrolling.
  This 13-item measure will be used to examine changes in caregiver knowledge, skill and confidence to manage their child. The PAM-DD also includes a rating scale of perceived caregiver activation level. The scale ranges from (1) strongly disagree to (4) strongly agree. A higher score indicates a more positive rating.
Parent Participation Engagement Measure | Measured at the completion of family navigation services for each family, approximately 4 months after enrolling.
  A 5-item parent-report measure of active caregiver engagement in youth mental health services. Each item assesses the frequency that a parent engaged in a participation behavior (e.g., asked questions, provided input, agreed with the plan) during a MH appointment on a 5-point scale ranging from (1) Not at all to (5) very much. To additionally capture family engagement, the investigators will track the number of contacts between the navigator and family during the interval between the PCP referral to navigation and the first completed MH appointment.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Broder-Fingert S, Stadnick NA, Hickey E, Goupil J, Diaz Lindhart Y, Feinberg E. Defining the core components of Family Navigation for autism spectrum disorder. Autism. 2020 Feb;24(2):526-530. doi: 10.1177/1362361319864079. Epub 2019 Jul 16. PMID 31311287
- [Background] Stadnick NA, Penalosa MG, Martinez K, Brookman-Frazee L, Gizzo DP, Sahms T, Kuelbs CL, Aarons GA. Pre-Implementation Organizational Environment Associated with Pediatric Integrated Care Readiness in Primary Care. Evid Based Pract Child Adolesc Ment Health. 2022;7(1):5-11. doi: 10.1080/23794925.2021.1875344. Epub 2021 Feb 5. PMID 35284636
- [Background] Stadnick NA, Martinez K, Aarons GA, Lee DA, Van Cleave J, Brookman-Frazee L. Pediatric Primary Care Perspectives on Integrated Mental Health Care for Autism. Acad Pediatr. 2020 Nov-Dec;20(8):1140-1147. doi: 10.1016/j.acap.2020.03.006. Epub 2020 Mar 20. PMID 32205263
- [Derived] Stadnick NA, Martinez K, Navarro F, Gomez-Patino P, Holmquist K, Negriff S, Roesch S, Bouchard I, Walpole S, Espinosa R, Broder-Fingert S, Barnett M, Brookman-Frazee L. Mixed Methods Findings from a Stepped Wedge Hybrid Implementation Trial of ATTAIN NAV: A Mental Health Family Navigation Intervention for Autistic Youth. J Autism Dev Disord. 2025 May 8. doi: 10.1007/s10803-025-06851-7. Online ahead of print. PMID 40338511